CLINICAL TRIAL: NCT02706327
Title: Comparison of Two Different Insole Types on Pain, Quality of Life and Physical Performance in Painful Flexible Flatfoot
Brief Title: Comparison of Two Different Insole Types in Painful Flexible Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasin YURT, Assist. Prof. Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/18-31
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Flatfoot
Keywords: orthotic insoles; pain; quality of life; athletic performance
MeSH Terms: conditions — Flatfoot; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAD/CAM (Experimental): 8-week follow-up with CAD/CAM insole and home based exercise program
  Interventions: Device: CAD/CAM Insole
- Semi-custom (Experimental): 8-week follow-up with semi-custom insole and home based exercise program
  Interventions: Device: Semi-custom Insole
- Control (Placebo Comparator): 8-week follow-up with placebo insole and home based exercise program
  Interventions: Other: Control

INTERVENTIONS:
Device: CAD/CAM Insole — A computer numerical control machine was used to product insoles according to pedobarographic pressure data;35 Shore A hardness ethyl vinyl acetate was used for the main insole, and 3 mm, 15 Shore A hardness ethyl vinyl acetate was used for covering. Orthotic insoles have been implemented in a pair of sports shoes.
  Arms: CAD/CAM
Device: Semi-custom Insole — Plantar surfaces of each patient's metatarsophalangeal joints were marked with a thick broad marker, and the participants were asked to stand on a clean paper. The borders of the foot were then drawn, and the medial longitudinal arch length was marked from the anterior aspect of the heel to the first metatarsophalangeal joint. These marks were used in designing and production. 35 Shore A hardness ethyl vinyl acetate was used for the main insole, and 3 mm, 15 Shore A hardness ethyl vinyl acetate was used for covering. Orthotic insoles have been implemented in a pair of sports shoes.
  Arms: Semi-custom
Other: Control — 15 Shore A hardness ethyl vinyl acetate, implemented in a pair of sports shoes as a placebo insole.
  Arms: Control

SUMMARY:
The purpose of this study is to compare computer aided design/computer aided manufacturing (CAD/CAM) and semi-custom insole types on pain, quality of life and physical performance and also to decide whether they are necessary in treatment of painful flexible flatfoot.

ELIGIBILITY:
Inclusion Criteria:

* minimum subtalar pronation of 5 degrees while standing (tibiocalcaneal angle, measured with goniometer),
* minimum of + 6 points on the foot posture index,

Exclusion Criteria:

* treatment of the foot for at least six months,
* leg length discrepancy of more than 1 cm,
* history of lower extremity surgery, and no disease that could affect lower extremity biomechanics.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Yurt, Dr., Principal Investigator — Eastern Mediterranean University

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between January 2014 and January 2016 at an outpatient clinic. Eligible participants were randomly assigned into three groups using simple randomization procedures.
Groups:
- CAD/CAM: 8-week follow-up with computer-aided design/computer aided manufacturing (CAD/CAM) insole and home based exercise program
  CAD/CAM Insole: A computer numerical control machine was used to product insoles according to pedobarographic pressure data;35 Shore A hardness ethyl vinyl acetate was used for the main insole, and 3 mm, 15 Shore A hardness ethyl vinyl acetate was used for covering. Orthotic insoles have been implemented in a pair of sports shoes.
Period: Overall Study
Arm/Group | CAD/CAM | Semi-custom | Control
Started | 22 | 22 | 23
Completed | 21 | 21 | 21
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAD/CAM | Semi-custom | Control | Total
Number analyzed (Participants) | 22 | 22 | 23 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.73 (2.89) | 23.05 (5.53) | 21.09 (1.95) | 21.94 (3.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 14 | 39
  Male | 9 | 10 | 9 | 28
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 23.03 (3.48) | 24.11 (4.15) | 23.32 (3.28) | 23.48 (3.62)
Foot Posture Index [Mean (Standard Deviation); unit: units on a scale] — This index measures posture (normal, pronated or supinated) of foot. Minimum-maximum values are -12 and +12 for the scale that 0 to +5 means normal foot posture, +6 to +9 means pronated foot, +10 and more means highly pronated and -1 to -4 means supinated foot, -5 to -12 means highly supinated.
  Subjects with +6 and more were participated in this study.
  units on a scale | 7.50 (1.73) | 8.59 (1.76) | 8.48 (2.04) | 8.19 (1.89)
Calcaneal valgus angle [Mean (Standard Deviation); unit: degree] | 6.36 (1.64) | 6.68 (1.67) | 6.22 (1.67) | 6.42 (1.65)
International Physical Activity Questionnaire Short Form [Mean (Standard Deviation); unit: kcal/week] | 3438.81 (3543.30) | 4731.27 (5392.45) | 2824.54 (2221.46) | 3688.98 (3389.92)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity Measured by 100 mm Visual Analog Scale
Description: The scale scores the pain intensity with 0 and 100 mm, minimum and maximum levels.
  Higher score means worse pain and also negative changes mean reduced pain. Participants were asked to rate the maximum level of foot pain they had in the last week.
  Changes were calculated as the difference between 8-week follow-up and baseline results.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: milimiters
Arm/Group | CAD/CAM | Semi-custom | Control
Number analyzed (Participants) | 22 | 22 | 23
milimiters | -31.40 (18.50) | -34.54 (14.24) | -12.08 (11.82)
Statistical Analysis 1: Comparison: CAD/CAM vs Semi-custom vs Control; Normality of the distribution was investigated by skewness-kurtosis, histogram graphics, normality tests and plots before the statistical tests were performed. Group comparisons were tested with One-way analysis of variance when normality was achieved and Kruskal Wallis test when not. A post-hoc test was used with Bonferroni correction; Test type: Other; p < 0.001, Kruskal-Wallis — A post-hoc test was used with Bonferroni correction and adjusted p-value was 0.016; Effect sizes (Cohen's d) were calculated for significant differences

2. Secondary Outcome: Change in Quality of Life Assessed With Short Form-36 Scale
Description: The scale scores the health related quality of life with 0 and 100, minimum and maximum levels.
  Each question is scored between 0-100 and the total score is found by dividing to number of question.
  Higher score or positive change mean better quality of life in the scale. We used physical health part of it.
  Changes were calculated as the difference between 8-week follow-up and baseline results.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAD/CAM | Semi-custom | Control
Number analyzed (Participants) | 22 | 22 | 23
units on a scale | 7.76 (11.04) | 6.68 (6.24) | 2.12 (4.75)
Statistical Analysis 1: Comparison: CAD/CAM vs Semi-custom vs Control; Normality of the distribution was investigated by skewness-kurtosis, histogram graphics, normality tests and plots before the statistical tests were performed. Group comparisons were tested with One-way analysis of variance when normality was achieved and Kruskal Wallis test when not; Test type: Other; p = 0.547, Kruskal-Wallis

3. Other Pre Specified Outcome: Balance Was Assessed With a Dynamic Platform
Description: Dynamic platform was the equipment used in balance assessment. Participants were assessed after using the insoles for 8 weeks in order to get compliance.
  Measurements were taken in the same day with and without insoles in shoes. The software calculates balance value between 0 and 5 that lower value means better balance score.
  Difference between with and without insole was calculated by subtracting the result with insole from the result without insole.
  Therefore, negative changes mean better balance score with insole.
Time Frame: In the same session after 8 weeks
Population: Two participants (1 CAD/CAM, 1 Semi-custom) did not bring their insole equipped shoes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAD/CAM | Semi-custom | Control
Number analyzed (Participants) | 20 | 20 | 21
units on a scale | -0.16 (0.77) | -0.29 (0.85) | -0.12 (1.08)
Statistical Analysis 1: Comparison: CAD/CAM vs Semi-custom vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.895, Kruskal-Wallis

4. Other Pre Specified Outcome: Six-minute Walk Physiological Cost Index Was Calculated
Description: Physiological cost index was calculated by taking heart rate with finger oximeter and walking distance after a six-minute walk test.
  The result is calculated by dividing one minute heart rate (beat) to walking distance (meter).
  Lower values mean better physiological cost. Participants were assessed after using the insoles for 8 weeks in order to get compliance.
  Measurements were taken in the same day with and without insoles in shoes. Difference between with and without insole was calculated by subtracting the result with insole from the result without insole.
  Therefore, negative changes mean better score with insole.
Time Frame: In the same session after 8 weeks
Population: Two participants (1 CAD/CAM, 1 Semi-custom) did not bring their insole equipped shoes.
Measure: Mean (Standard Deviation); unit: beat/meter
Arm/Group | CAD/CAM | Semi-custom | Control
Number analyzed (Participants) | 20 | 20 | 21
beat/meter | 0.017 (0.12) | 0.007 (0.09) | 0.029 (0.16)
Statistical Analysis 1: Comparison: CAD/CAM vs Semi-custom vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.842, Kruskal-Wallis

5. Other Pre Specified Outcome: Vertical Jump Height Was Measured With a Special Mat
Description: Sensor mat was used in vertical jump measurement. The result is the distance (cm) that was jumped vertically and it is normalized by dividing the distance to length of subject in order to get percentage of jump distance.
  Higher values mean better vertical jump performance. Participants were assessed after using the insoles for 8 weeks in order to get compliance.
  Measurements were taken in the same day with and without insoles in shoes. Difference between with and without insole was calculated by subtracting the result with insole from the result without insole.
  Therefore, positive changes mean better score with insole.
Time Frame: In the same session after 8 weeks
Population: Two participants (1 CAD/CAM, 1 Semi-custom) did not bring their insole equipped shoes.
Measure: Mean (Standard Deviation); unit: percentage of distance
Arm/Group | CAD/CAM | Semi-custom | Control
Number analyzed (Participants) | 20 | 20 | 21
percentage of distance | 0.35 (0.85) | 0.19 (0.95) | 0.87 (1.38)
Statistical Analysis 1: Comparison: CAD/CAM vs Semi-custom vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.848, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Through 8-week follow up period.
Description: Deteriorating of foot pain was defined as a potential adverse event of insole and measured by using (0-100 mm) visual analog scale, that higher means worse, at the time subject was reported the event.
Arm/Group | CAD/CAM | Semi-custom | Control
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAD/CAM (N=22) | Semi-custom (N=22) | Control (N=23)
Increase in foot pain during follow up period. (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Subjects were asked to report if their foot pain got worse at any time.

LIMITATIONS AND CAVEATS:
The young average age of our study population could limit the generalizability of our results and the two-month follow-up interval was sufficient to see the benefit of insoles but may not be long enough to determine whether the benefit will last.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No